CLINICAL TRIAL: NCT05417724
Title: Utilizing Battlefield Acupuncture(BFA) to Treat Chronic Pain for Homeless and at Risk Veterans.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edith Nourse Rogers Memorial Veterans Hospital (U.S. Federal Agency)
Responsible Party: Principal Investigator, Cathy St. Pierre, Principal Investigator, Edith Nourse Rogers Memorial Veterans Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1645513
Record Dates: First submitted 2022-05-19; First posted 2022-06-14 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Acupuncture; Homelessness; Pain; Veterans
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Recruitment of veterans with chronic pain who are interested in being treated with Battlefield Acupuncture (BFA).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Battlefield Acupuncture (Other): All subjects will receive BFA treatment weekly for 12 weeks.
  Interventions: Other: Battlefield Acupuncture

INTERVENTIONS:
Other: Battlefield Acupuncture — Battlefield Acupuncture

SUMMARY:
This research study will evaluate the effectiveness of utilizing Battlefield Acupuncture (BFA) on homeless and at risk for homelessness veterans with chronic pain for 12 weeks.

DETAILED DESCRIPTION:
Methodology: This is a mixed methods prospective design study. A total of 35 subjects will be recruited for this study. The primary study outcome variables are: pain level- pre and post treatment, stress, mood and usual activity levels, sleep patterns and behavioral factors such as ; anxiety, depression, suicidal ideation, substance use and housing stability.

4. Findings: Pending

5. Clinical Relationships: This study is conducted to demonstrate whether or not BFA treatment will decrease pain and improve quality of life for homeless and at risk for homelessness veterans.

6. Impact/Significance: Pending

ELIGIBILITY:
Inclusion Criteria:

Eligibility criteria include:

* they are 18 years or older
* they are homeless or at risk for homelessness veterans who are enrolled in the VA Bedford Healthcare system and registered in one of the HUD-VASH or HCHV programs,
* history of chronic pain.
* Availability to participate in the study for 4 months.

If they meet these criteria, they will be asked to complete the Informed consent to enroll in the study.

Exclusion Criteria:

* female veterans who are pregnant
* history of bleeding disorders or currently on blood thinning medications
* currently being treated for an active infection of the outer ear.
* currently have a PICC line in their body or are receiving IV antibiotics.
* fear of needles/tacks
* undiagnosed pain complaint

Our recruitment plan invites all eligible veterans and is just, fair, and equitable.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2023-09-05 (Actual); Study Completion 2023-09-05 (Actual)

PRIMARY OUTCOMES:
Reduction in pain | 4 months
  Whether the use of BFA on veterans with chronic pain will decrease pain. Questionnaire. The pain scale is based on 0-10 with a higher score indicating an increase in pain and the lower score indicating a decrease in pain level.

SECONDARY OUTCOMES:
Change in pain may impact behavioral health issues. | 4 months
  Whether effective treatment for chronic pain has an impact on behavioral health issues. Patient Health Questionnaire (PHQ-4) will measure changes in anxiety and depression based on a numerical score from 0-4. This questionnaire is broken down into 4 questions- 2 focused on anxiety and two questions focused on depressions. Each question has a likert scale to select a number from 0-3. The higher the number, the higher the level of anxiety/depression. The cumulative score is based on a score of 0-12, with the higher scores indicating higher psychological distress.
Change in pain may impact housing stability | 4 months
  Whether effective treatment for chronic pain has an impact on housing stability as measured by the housing stability questionnaire. this questionnaire asks questions about the number of nites in the past 30 days, a research subject has spent in a variety of settings. The scale is 0-30 with the higher the number, the more transient the person's current living situation. The purpose is to see if a change in pain levels will impact the number of nights in transitional housing. The higher the pain level an positively/negatively impact the numbers of nite in transitional housing
Change in pain may impact substance use. | 4 months
  Whether effective treatment for chronic pain has an impact on substance use as measured by the substance use questionnaire. This questionnaire asked each subject to identify the number of drinks/drugs that the subject has consumed in the past 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: John Wells, PhD, Study Chair — Edith Nourse Rogers Memorial Veterans Hospital
Locations (1):
- Bedford VA Healthcare System, Bedford, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
No plan to do this.

DOCUMENTS (1):
  • Informed Consent Form (2022-09-19): https://cdn.clinicaltrials.gov/large-docs/24/NCT05417724/ICF_000.pdf